CLINICAL TRIAL: NCT02648737
Title: Cognitive Behavioural Therapy for Anxiety Disorders in Patients With Parkinson's Disease: a Randomized, Controlled Trial of the Clinical Effectiveness and Changes in Cerebral Connectivity
Brief Title: Cognitive Behavioural Therapy for Anxiety Disorders in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Anja Moonen, post doctoral researcher, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11169
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Parkinson's Disease; Generalized Anxiety Disorder; Social Phobia
Keywords: Parkinson's disease; Cognitive Behavioural therapy; generalized anxiety disorder; social phobia; cerebral connectivity
MeSH Terms: conditions — Parkinson Disease; Generalized Anxiety Disorder; Phobia, Social | interventions — Cognitive Behavioral Therapy; Clinical Trials Data Monitoring Committees

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioural Therapy (CBT) (Experimental): Patients who will receive CBT plus clinical monitoring will receive 10 weekly individual sessions (60-75 minutes), tailored to the preferences and needs of each patient. In each session, a registered psychologist will address specified aspects of (coping with) anxiety and related concerns with a specific focus on behaviour and thoughts associated with anxiety.
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT); Other: Clinical monitoring
- Clinical monitoring (Other): Patients assigned to clinical monitoring only will receive general education material on coping with PD symptoms and behavioural symptoms such as anxiety. In addition, they will be followed-up 1 month after baseline assessment via telephone calls to inquire about current anxiety symptoms. Patients will remain under the care of their personal physicians, who will also monitor their medical and psychiatric status. Patients who receive clinical monitoring only will be given the option to receive CBT once the trial is completed.
  Interventions: Other: Clinical monitoring

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT) — Cognitive Behavioural Therapy (CBT) is considered the gold standard in psychotherapeutic treatments of anxiety. CBT is defined as: 'An amalgam of behavioural and cognitive problem-based interventions guided by principles of applied science. The behavioural interventions aim to decrease maladaptive behaviours and increase adaptive ones by modifying their antecedents and consequences and by behavioural practices that result in new learning. The cognitive interventions aim to modify maladaptive cognitions, self-statements, or beliefs.' (Arch & Craske, 2009; Craske, 2010).
  Arms: Cognitive Behavioural Therapy (CBT)
Other: Clinical monitoring — Patients assigned to clinical monitoring only will receive general education material on coping with PD symptoms and behavioural symptoms such as anxiety. In addition, they will be followed-up 1 month after baseline assessment via telephone calls to inquire about current anxiety symptoms. Patients will remain under the care of their personal physicians, who will also monitor their medical and psychiatric status.

SUMMARY:
Anxiety disorders occur in up to 35% of patients with Parkinson's disease (PD) and have a negative effect on gait, dyskinesia, freezing, on/off fluctuations, and quality of life. With this Randomized Controlled Trial the investigators intend to 1) develop a Cognitive Behavioural Therapy (CBT) module for anxiety in PD 2) assess the effectiveness of this module in reducing anxiety symptoms, and 3) study the effects of CBT on cerebral connectivity. Effective CBT treatment of anxiety will provide patients with behavioural and anxiety management techniques that can give lasting benefits, not only on anxiety symptoms, but potentially also on motor symptoms.

DETAILED DESCRIPTION:
Anxiety is common in patients with Parkinson's disease (PD) and has a negative effect on several motor symptoms and quality of life in general. So far, there is no treatment, neither pharmacological nor psychotherapeutic, that intends to specifically reduce anxiety symptoms in PD. Cognitive Behavioural Therapy (CBT) is an effective treatment for anxiety disorders in patients without PD. In PD, CBT is an effective treatment for depression and for impulse control disorders (ICD). PD patients who received CBT for depression reported not only a reduction in depression and comorbid anxiety, but also a beneficial influence on coping and quality of life, compared to PD patients who only received clinical monitoring. In addition to the clinical effectiveness, several studies have demonstrated the therapeutic effects of CBT on functional neural activity. The two most common anxiety disorders in patients with Parkinson's Disease (PD): generalized anxiety disorder (GAD) and social anxiety disorder (SAD) are both characterized by dysfunctional connectivity between limbic areas (among which the amygdala) and the frontal cortex. Recent functional imaging studies have shown that CBT can alter neural correlates of affective processing by increasing functional connectivity between limbic and frontal cortices. The present study aims to study the clinical effectiveness of a CBT module for the treatment of the two most common anxiety disorders in patients with Parkinson's Disease (PD): generalized anxiety disorder (GAD) and social anxiety disorder (SAD) in a randomized controlled trial (RCT). The CBT module will be based on existing modules for anxiety disorders in non-PD patients, and on modules for depression and ICD in PD patients. In addition, the investigators aim to get more insight into biological dysfunction associated with anxiety in PD, as well as alterations in brain structure, brain function and cerebral connectivity due to CBT. The investigators will study the biological correlates of successful treatment by using structural and functional magnetic resonance-imaging (MRI) scanning. The present study further aims to study the long term clinical effectiveness of the CBT module, measured by the change anxiety score after 3 and 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD according to the Queens Square Brain Bank diagnostic criteria
* Presence of clinically relevant anxiety symptoms, as operationalized by the Mini International Neuropsychiatric Inventory (MINI), sections for social phobia (F) and GAD (H), and/or a Parkinson Anxiety Scale (PAS) persistent score >9 and/or PAS avoidance score >3.
* Using a stable dose of levodopa or other antiparkinsonian medication for at least one month
* No other current psychological treatment for anxiety; pharmacotherapy (e.g., selective serotonin re-uptake inhibitors) is allowed if a stable dose is used at least 2 months prior to participation and the patient still meets inclusion criteria. During the trial the dosage should not be changed. Medication use and mental health care will be tracked throughout the study.
* Signed informed consent

Note: In order to achieve a representative study sample, patients will be included irrespective of their disease stage or their current antiparkinsonian medication.

Exclusion Criteria:

* Parkinsonian syndromes or neurodegenerative disorders other than PD
* Dementia or severe cognitive decline, operationalized as a Montreal Cognitive Assessment (MOCA) score < 24
* Contra-indications for magnetic resonance imaging
* Major depressive disorder (MDD) as defined by the criteria of a DSM-V diagnosis for MDD
* Abuse of alcohol, drugs or benzodiazepines.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change in anxiety score as measured with the Hamilton Anxiety Rating Scale (HARS). | Baseline assessment (T0) and post-treatment assessment (T1; after 10 weeks)

SECONDARY OUTCOMES:
Changes in cerebral connectivity between limbic and frontal cortices as measured with resting state blood-oxygen-level dependent functional magnetic resonance imaging (BOLD fMRI) and diffusion tensor imaging (DTI) | MRI scanning at baseline (T0) and post-treatment (T1; after 10 weeks)
Long term clinical effectiveness of the CBT module measured by the change in HARS score | 3 months follow-up (T2) and 6 months follow-up (T3)

CONTACTS AND LOCATIONS:
Overall Officials: Albert FG Leentjens, MD, PhD, Study Director — Maastricht University Medical Centre
Locations (2):
- Neurology and Movement Disorders Unit, Lille University Hospital, Lille, France
- Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Treatment module will be made available for public use. Study data will be published in peer-reviewed journals.

REFERENCES:
- [Derived] Mulders AEP, Moonen AJH, Dujardin K, Kuijf ML, Duits A, Flinois B, Handels RLH, Lopes R, Leentjens AFG. Cognitive behavioural therapy for anxiety disorders in Parkinson's disease: Design of a randomised controlled trial to assess clinical effectiveness and changes in cerebral connectivity. J Psychosom Res. 2018 Sep;112:32-39. doi: 10.1016/j.jpsychores.2018.04.002. Epub 2018 Apr 10. PMID 30097133